CLINICAL TRIAL: NCT07176390
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tulisokibart in Participants With Rheumatoid Arthritis
Brief Title: A Clinical Study of Tulisokibart (MK-7240) to Treat Rheumatoid Arthritis (RA) (MK-7240-014)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7240-014; U1111-1320-8718 (Registry Identifier: UTN); 2025-521745-25-00 (Registry Identifier: EU CT); MK-7240-014 (Other: MSD)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High-dose tulisokibart (Experimental): Participants receive background therapy of methotrexate (MTX) PLUS a high dose of tulisokibart
  Interventions: Drug: Tulisokibart; Drug: Methotrexate
- Medium-dose tulisokibart (Experimental): Participants receive background therapy of MTX PLUS a medium dose of tulisokibart.
  Interventions: Drug: Tulisokibart; Drug: Methotrexate
- Low-dose tulisokibart (Experimental): Participants receive background therapy of MTX PLUS a low dose of tulisokibart and are rerandomized at week 12 to a medium or high dose of tulisokibart.
  Interventions: Drug: Tulisokibart; Drug: Methotrexate
- Placebo (Placebo Comparator): Participants receive background therapy of MTX PLUS a dose-matched tulisokibart placebo and are re-randomized at week 12 to a medium or high dose of tulisokibart.
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: Tulisokibart — Subcutaneous (SC) administration
  Other Names: MK-7240; PRA023
  Arms: High-dose tulisokibart; Low-dose tulisokibart; Medium-dose tulisokibart
Drug: Placebo — SC Injection
  Arms: Placebo
Drug: Methotrexate — Background Therapy - SC injection or oral administration. Per protocol, parenteral administration is allowed.
  Other Names: MTX

SUMMARY:
Researchers are looking for new ways to treat rheumatoid arthritis (RA). Methotrexate (MTX) is a standard (usual) treatment for RA. However, MTX and other current treatments may not work well to treat RA symptoms for many people.

This study will help find out if a study medicine called tulisokibart can treat symptoms of active RA in people who are taking MTX. In this study, researchers will look at different doses of tulisokibart.

Researchers want to learn if at least one of the study doses of tulisokibart works better than a placebo to lessen RA symptoms. A placebo looks like the study medicine but has no study medicine in it. Using a placebo helps researchers better understand the effects of the study medicine.

DETAILED DESCRIPTION:
This study consists of a 12-week Placebo-controlled Period and a 116-week Long-term Extension (LTE), which is composed of a 44-week Main Extension and an 72-week Optional Extension

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a clinical diagnosis of rheumatoid arthritis (RA) and fulfillment of 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria
* Has active disease defined as ≥6 tender joints (based on 68 joints) and ≥6 swollen joints (based on 66 joints)
* Has current treatment with oral or parenteral methotrexate (MTX) therapy
* Has history of one of the following: a) biologic disease-modifying antirheumatic drug (bDMARD) naïve, or b) bDMARD-Inadequate Response (IR)/intolerant up to a maximum of 2 classes of bDMARDS

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has any arthritis with onset before age 17 years or current diagnosis of inflammatory joint disease other than RA (such as, but not limited to, psoriatic arthritis, systemic lupus erythematosus, gout, systemic sclerosis, myositis, pseudogout, etc) or any other condition that may, in the judgment of the investigator, interfere with the assessment of RA
* Has a history of cancer (except fully treated nonmelanoma skin cancers or cervical carcinoma in situ after complete surgical removal) and is disease free for <5 years before randomization
* Has any active infection
* Has known allergies, hypersensitivity, or intolerance to tulisokibart or its excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-03-08 (Estimated); Study Completion 2029-09-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving American College of Rheumatology 20% Response Criteria (ACR20) at Week 12 | Week 12
  The ACR20 response is a composite measure to evaluate disease activity in RA. ACR20 response is defined as a ≥20% improvement in: a) swollen joint count (66 joints) and tender joint count (68 joints) (0= Absent; 1= Present) and b) ≥20% improvement in ≥3 of the following 5 assessments and questionnaires: i) Health Assessment Questionnaire Disability Index (HAQ-DI) (0=without any difficulty; 3= unable to do) a higher score=worse disability, ii) Physician Global Assessment of Disease Activity (PGA) (0= not active to 10= very active) a higher score= more active disease; iii) Patient's Global Assessment of Disease Activity (PtGA) (0= not active to 10= very active) a higher score= more active disease; iv) Patient assessment of Pain Severity (0= no pain to 10= most severe pain) a higher score = more pain; v) High-sensitivity C-reactive protein (hsCRP) serum values, a lower value indicates less inflammation. The proportion of participants with ACR20 response at Week 12 will be presented.

SECONDARY OUTCOMES:
Proportion of Participants Achieving American College of Rheumatology 50% Response Criteria (ACR50) at Week 12 | Week 12
  The ACR50 response is a composite measure to evaluate disease activity in RA. ACR50 response is defined as a ≥50% improvement in: a) swollen joint count (66 joints) and tender joint count (68 joints) (0= Absent; 1= Present) and b) ≥50% improvement in ≥3 of the following 5 assessments and questionnaires: i) Health Assessment Questionnaire Disability Index (HAQ-DI) (0= without any difficulty; 3= unable to do) a higher score=worse disability, ii) Physician Global Assessment of Disease Activity (PGA) (0= not active to 10= very active) a higher score= more active disease; iii) Patient's Global Assessment of Disease Activity (PtGA) (0= not active to 10= very active) a higher score= more active disease; iv) Patient assessment of Pain Severity (0= no pain to 10= most severe pain) a higher score = more pain; v) High-sensitivity C-reactive protein (hsCRP) serum values, a lower value indicates less inflammation. The proportion of participants with ACR50 response at Week 12 will be presented.
Proportion of Participants Achieving American College of Rheumatology 70% Response Criteria (ACR70) at Week 12 | Week 12
  The ACR70 response is a composite measure to evaluate disease activity in RA. ACR70 response is defined as a ≥70% improvement in: a) swollen joint count (66 joints) and tender joint count (68 joints) (0= Absent; 1= Present) and b) ≥70% improvement in ≥3 of the following 5 assessments and questionnaires: i) Health Assessment Questionnaire Disability Index (HAQ-DI) (0= without any difficulty; 3= unable to do) a higher score=worse disability, ii) Physician Global Assessment of Disease Activity (PGA) (0= not active to 10= very active) a higher score= more active disease; iii) Patient's Global Assessment of Disease Activity (PtGA) (0= not active to 10= very active) a higher score= more active disease; iv) Patient assessment of Pain Severity (0= no pain to 10= most severe pain) a higher score = more pain; v) High-sensitivity C-reactive protein (hsCRP) serum values, a lower value indicates less inflammation. The proportion of participants with ACR70 response at Week 12 will be presented.
Proportion of Participants Achieving Low Disease Activity (LDA) based on Disease Activity Score 28 Using C-Reactive Protein (DAS28-CRP) | Week 12
  The DAS28-CRP is a composite measure of RA disease activity. DAS28-CRP is based upon a statistically-derived index combining the following 4 components: i) tender joint count (TJC) (28 joints; 0=absent, 1=present; TJC28), ii) swollen joint count (SJC) (28 joints; 0=absent, 1=present; SJC28), iii) serum high-sensitivity C-reactive protein (hsCRP), serum value decrease indicates less inflammation, and iv) Patient's Global Assessment of Disease Activity (PtGA) (0= not active to 10= very active) a higher score= more active disease. The index is defined as follows: DAS28-CRP = 0.56 × SQRT(TJC28) + 0.28 × SQRT(SJC28) + 0.36 × ln (hsCRP+1) + 0.014 × ptGA+ 0.96. The DAS28-CRP is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. Remission is indicated by a DAS28-CRP score of <2.6 and low disease activity (LDA) by a DAS28-CRP score of ≤3.2. The proportion of participants who achieve LDA will be presented.
Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 12 | Baseline and Week 12
  The HAQ-DI is a 20-item questionnaire that measures physical function in participants with RA. The questionnaire assesses the degree of difficulty a person has in accomplishing tasks in 8 functional area domains (dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area domain are scored from 0 to 3 (0= without any difficulty; 3= unable to do), with a higher score indicating inability to perform activity. The overall disability score (HAQ-DI) is a summation of the highest score from each domain divided by the number of domains completed and ranges from 0 to 3, with the higher value indicating worse disability. The change from baseline to week 12 in the HAQ-DI score will be presented.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately Week 142
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately Week 128
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (55):
- United States (16):
  - Arizona Arthritis & Rheumatology Associates, P.C. ( Site 1018), Glendale, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Mesa ( Site 1033), Mesa, Arizona
  - Arthritis & Osteoporosis Medical Center - La Palma ( Site 1024), La Palma, California
  - Tekton Research, LLC. ( Site 1008), Fort Collins, Colorado
  - Sweet Hope Research Specialty, Inc ( Site 1015), Hialeah, Florida
  - HMD Research LLC ( Site 1016), Orlando, Florida
  - Greater Chicago Specialty Physicians - Orland Park ( Site 1043), Orland Park, Illinois
  - AA Medical Research Center ( Site 1027), Grand Blanc, Michigan
  - Kansas City Physician Partners ( Site 1032), Kansas City, Missouri
  - Physician Research Collaboration, LLC ( Site 1002), Lincoln, Nebraska
  - altoona center for clinical research ( Site 1005), Duncansville, Pennsylvania
  - Rheumatology Specialty Center ( Site 1030), Willow Grove, Pennsylvania
  - AARA Clinical Research - Murfreesboro Medical Clinic ( Site 1034), Murfreesboro, Tennessee
  - Rheumatology Associates ( Site 1026), Arlington, Texas
  - Epic Medical Research ( Site 1004), Red Oak, Texas
  - Advanced Rheumatology of Houston - Woodlands ( Site 1000), The Woodlands, Texas
- Canada (2):
  - CIUSSS de l'Estrie - CHUS, Hotel-Dieu de Sherbrooke ( Site 1106), Sherbrooke, Quebec
  - Centre de Recherche Musculo-Squelettique ( Site 1101), Trois-Rivières, Quebec
- China (7):
  - Peking University First Hospital ( Site 2511), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University. ( Site 2510), Xiamen, Fujian
  - The Third Affiliated Hospital, Sun Yat-sen University ( Site 2514), Guangzhou, Guangdong
  - Xinxiang Central Hospital ( Site 2501), Xinxiang, Henan
  - Linfen Central Hospital ( Site 2507), Linfen, Shanxi
  - PEOPLE'S HOSPITAL OF XINJIANG UYGUR AUTONOMOUS REGION ( Site 2515), Ürümqi, Xinjiang
  - Taizhou Hospital of Zhejiang Province ( Site 2506), Linhai, Zhejiang
- Colombia (3):
  - Clinica de la Costa S.A.S. ( Site 1301), Barranquilla, Atlántico
  - CIREEM SAS ( Site 1304), Bogota, Cundinamarca
  - Fundación Valle del Lili ( Site 1305), Cali, Valle del Cauca Department
- Germany (4):
  - Medicover München Ost MVZ ( Site 1607), München, Bavaria
  - Rheuma-Research Lausitz ( Site 1604), Cottbus, Brandenburg
  - Rheumatologische Schwerpunktpraxis ( Site 1603), Berlin
  - HRF II - Hamburger Rheuma Forschungszentrum II MVZ für Rheumatologie und Autoimmunmedizin Hamburg G ( Site 1602), Hamburg
- Japan (6):
  - Toshin Yoshida Internal Medicine Rheumatology ( Site 2606), Hanishina-gun, Nagano
  - Sasebo Chuo Hospital ( Site 2602), Sasebo, Nagasaki
  - Nagaoka Red Cross Hospital ( Site 2604), Nagaoka, Niigata
  - Hirose Clinic ( Site 2601), Tokorozawa, Saitama
  - University of Yamanashi Hospital ( Site 2603), Chūō, Yamanashi
  - Kai Clinic ( Site 2600), Miyazaki
- Poland (7):
  - MICS Centrum Medyczne Bydgoszcz ( Site 1807), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki nr 2 im. Dr. Jana Biziela-Klnk Reumatologii i Ukladowych Chorob Tkanki Lacznej ( Site 1804), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun ( Site 1803), Torun, Kuyavian-Pomeranian Voivodeship
  - Zespół Poradni Specjalistycznych Reumed Filia nr 1 Wallenroda ( Site 1801), Lublin, Lublin Voivodeship
  - MICS Centrum Medyczne Warszawa ( Site 1805), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji ( Site 1806), Warsaw, Masovian Voivodeship
  - NZOZ BIF-MED ( Site 1802), Bytom, Silesian Voivodeship
- South Korea (3):
  - Soon Chun Hyang University Cheonan Hospital ( Site 2304), Cheonan-si, Chungcheongnam-do
  - Chungnam national university hospital ( Site 2303), Daejeon, Taejon-Kwangyokshi
  - Hanyang University Seoul Hospital ( Site 2300), Seoul
- Spain (4):
  - Hospital Universitari Parc Tauli ( Site 1900), Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla ( Site 1906), Santander, Cantabria
  - Hospital Clinico Universitario de Santiago ( Site 1903), Santiago de Compostela, La Coruna
  - Hospital Universitari Vall d'Hebron ( Site 1901), Barcelona
- United Kingdom (3):
  - The Princess Alexandra Hospital NHS Trust ( Site 2103), Harlow, England
  - Chapel Allerton Hospital ( Site 2106), Leeds
  - Barnet Hospital ( Site 2102), London

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com